CLINICAL TRIAL: NCT05189535
Title: "Evaluation of the Effect of Pentoxifylline on the Prevention of Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients"
Brief Title: "Prevention of Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients"
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sondos Sherif Ismail, Clinical Pharmacy, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: s2192648
Record Dates: First submitted 2021-10-04; First posted 2022-01-12 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Female; Peripheral Neuropathy
Keywords: Breast cancer; pentoxifylline; paclitaxel; Taxol; peripheral neuropathy; Trental
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Pentoxifylline; Paclitaxel

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, placebo controlled
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pentoxifylline 400 mg (Experimental): Patients will receive paclitaxel 80 mg/m2 once per week for 12 weeks and pentoxifylline 400 mg twice daily for the paclitaxel treatment period.
  Interventions: Drug: Pentoxifylline; Drug: Paclitaxel
- Placebo (Placebo Comparator): Patients will receive paclitaxel 80 mg/m2 once per week for 12 weeks and placebo twice daily for the paclitaxel treatment period..
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400 mg oral tablet twice daily for 12 weeks.
  Other Names: Trental
  Arms: pentoxifylline 400 mg
Drug: Paclitaxel — Paclitaxel I.V 80 mg/m2 weekly
  Other Names: Taxol
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effect of pentoxifylline 400 mg twice daily administration on the prevention of paclitaxel-Induced peripheral neuropathy in breast cancer patients.

DETAILED DESCRIPTION:
Paclitaxel induced peripheral neuropathy (PIPN) starts early during therapy and may worsen even after cessation and affect mainly sensory neurons. The symptoms of neuropathy include pain, tingling, cold-sensitivity and numbness that typically presents in a stocking glove distribution. The pathogenesis of PIPN may be attributed to drug accumulation in dorsal root ganglia causing increase in inflammatory cytokines, immune mediators and dysregulation of calcium subunits which in turn increases pain. It also causes oxidative stress in sensory axons leading to axon demyelination, increased sensitization to signal transduction, release of pro-inflammatory mediators and activation of apoptosis.

Many animal studies and clinical trials have shown pentoxifylline to have a significant anti-inflammatory and antioxidant effect. It also preserved nerve conduction velocity and ameliorated mechanical hyperalgesia. Pentoxifylline showed a prominent reduction in neuropathic pain in diabetic patients. These effects were mainly due to the ability of pentoxifylline to reduce TNF-α and MDA levels. So, pentoxifylline is a drug of interest due to its ability to ameliorate neuro-inflammation and oxidative stress which play a critical role in PIPN pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-80 years old).
* Female patients.
* Pathologically proved breast cancer.
* Breast cancer patients who will receive adjuvant and neoadjuvant weekly paclitaxel for 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance ≤ 2
* Adequate bone marrow function.
* Adequate liver and kidney function.

Exclusion Criteria:

* Patients with preexisting clinical neuropathy.
* Patients with diabetes mellitus.
* Metastatic breast cancer.
* Patients receiving medications that ameliorate neuropathy like; antidepressants, anticonvulsants, opioids, adjuvant or topical analgesics.
* Patients treated with medications that increase the risk of neuropathy.
* Hypersensitivity to pentoxifylline or xanthine derivatives.
* Patients with recent (within 1 month) surgery, myocardial infarction (MI), intracranial or retinal bleeding or active peptic ulcer.
* Patients at high risk for bleeding or taking medications that increase risk of bleeding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Paclitaxel induced-peripheral neuropathy | 12 weeks
  Number of patients reported neuropathy due to paclitaxel

SECONDARY OUTCOMES:
Grade of severity of Paclitaxel induced-peripheral neuropathy in patients who developed neuropathy | at baseline and on weekly bases for 12 weeks
  Severity of neuropathic symptoms will be graded using Common Terminology Criteria for Adverse Events Version 5 (CTCAE v5)
Evaluation of Safety and tolerability of pentoxifylline | evaluation on weekly bases for 12 weeks.
  side effects reported due to pentoxifylline will be recorded.
The need for dose reduction or drug discontinuation in pentoxifylline and placebo arm. | 12 weeks
  number of patients who needed dose reduction or drug discontinuation due to paclitaxel induced neuropathy will be recorded.

OTHER OUTCOMES:
Serum tumor necrosis factor alpha (TNF-α) | at baseline and after 12 weeks
  measuring serum level of tumor necrosis factor using ELISA kit
Serum malondialdehyde (MDA) | at baseline and after 12 weeks
  measuring serum level of malondialdehyde.
The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity(FACT-GOG-NTX) subscale | at baseline, week 1 in each cycle (cycle length is 21 days) up to 12 weeks and at week 12.
  evaluating the functional difficulties and quality of life related to paclitaxel induced neuropathic symptoms.
  score range from (0-44) where lower score indicates more sever symptoms according to the FACT-GOG-NTX scoring guideline.
Time to develop neuropathy | 12 weeks
  mean time to develop grade 3 or 4 neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No